CLINICAL TRIAL: NCT04786288
Title: The Effect of Aromatherapy Hand Massage on Pain Level and Vital Signs in Elderly People With Chronic Non-malignant Pain
Brief Title: Reliving Chronic Non-malignant Pain of Elderly Individuals Using Aromatic Hand Massage
Acronym: RCNMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haben Tesfu Gebreselassie (Other)
Responsible Party: Sponsor-Investigator, Haben Tesfu Gebreselassie, Sponsor-Investigator, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19-4.1T/26
Record Dates: First submitted 2021-02-28; First posted 2021-03-08 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Non-malignant Chronic Pain
Keywords: aromatherapy; elderly; massage; pain; vital signs
MeSH Terms: conditions — Pain | interventions — Massage

STUDY DESIGN:
Intervention Model Description: simple and stratified randomization method (experiment, control and placebo group x pre-test post-test)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aromatherapy (Experimental): 22 elderly participants received M technique hand massage that lasted for 10 minutes for both their hands and arms using 2% lavender essential oil diluted with odourless baby oil (12 drops of lavender essential oil mixed in 30 ml of carrier oil) was used to apply the hand massage.
  Intervention: massage with lavender essential oil mixed in a carrier oil
  Interventions: Other: massage with lavender essential oil mixed in a carrier oil
- Placebo (Placebo Comparator): odourless baby oil was used for the application of the M technique hand massage on both hands and arms for 10 minutes for the 22 elderly participants.
  Intervention: other: massage with no fragrance baby oil
  Interventions: Other: massage with odourless baby oil
- Control (No Intervention): Participants in this group didn't receive any type of intervention from the researcher except the routine hospital management.

INTERVENTIONS:
Other: massage with lavender essential oil mixed in a carrier oil — 22 elderly participants received a one session M technique hand massage that lasted 10 minutes for both their hands and arms using 2% lavender essential oil diluted with odourless baby oil (12 drops of lavender essential oil mixed in 30 ml of carrier oil) was used to apply the M technique hand massage
  Arms: Aromatherapy
Other: massage with odourless baby oil — odourless baby oil was used for the application of one session M technique hand massage on both hands and arms for 10 minutes for the 22 elderly participants.
  Arms: Placebo

SUMMARY:
This randomized controlled study was conducted to determine the effect of hand aromatherapy massage on non-malignant chronic pain.

Total of 66 elderly individuals who had visited an algology outpatient polyclinic with a complaint of chronic non-malignant pain for at least three months were randomly assigned to the study. Participants were allocated to three groups and aromatherapy massage was done for those in the intervention group while odourless baby oil was used during the hand massage in the placebo group, those participants in the control group did not receive any type of intervention. Data collection was carried out using Individual Diagnosis Form, Visual Analogue Scale and Brief Pain Inventory. Before and after intervention, data collection forms were filled and pain level and vital signs were evaluated.

Participants pain severity after aromatherapy decreased by 42.24%. When comparing vital sign pre-post procedure; systolic blood pressure value for the placebo group was significantly lower. Right after intervention, pulse rate was significantly lower in aromatherapy and placebo groups while post intervention body temperature in aromatherapy group was found to be higher and statistically significant.

This study has shown that aromatherapy hand massage is effective on lowering pain level and positively influencing vital signs of elderly individuals with chronic non-malignant pain. Considering these beneficial effects, aromatherapy massage can be used as an independent nursing intervention in elderly individuals who are suffering from chronic pain.

DETAILED DESCRIPTION:
This research study was designed as a randomized placebo-controlled clinical trial to examine the effect of aromatherapy hand massage on chronic non-malignant pain and vital signs of elderly individuals. Sample size was determined via G-power statistical analysis with 95% conﬁdence and 80% theoretical power. Initially pilot study was performed with total of 6 elderly patients, 2 individuals for each group. Those elderly patients who visited the polyclinic on Monday were appointed to aromatherapy group (n=22), those who came on Wednesday they were assigned to placebo group (n=22) and those who visited the clinic on Friday were allocated to control group (n=22). Individuals who were included in this research were age 65 and above, must have chronic non-malignant pain for at least three months, should not have cognitive impairment, must be able to answer questions independently and those who have agreed to be part of the study were included in the sample. In the contrary, patients with dermatological problems, swelling, sign of inflammation, neuropathy or loss of sensation and deformity on their hands and/ or arms were excluded from the study and cancer patients and those who had allergic to lavender oil were also excluded.

Data were gathered as patient information form, visual analogue scale (VAS), brief pain inventory and vital signs which were collected by a single researcher via face-to-face interview and hand massage was performed by the same researcher.

In the aromatherapy group written and verbal consent was obtained from participants prior the intervention after that patient information form was filled, pain level was assessed via visual analogue scale (VAS) and brief pain inventory, vital signs were assessed as well. M technique hand massage was done on both hands and arms for 10 minutes using lavender essential oil (12 drops of lavender essential oil mixed in 30 ml of fragrance-free baby oil as a carrier oil) afterwards pain level was re-assessed using usual analogue scale and vital signs were re-evaluated within 10-15 minutes after the completion of the intervention.

In the placebo group written and verbal consent was obtained from participants prior the intervention after that patient information form was filled, pain level was assessed via visual analogue scale (VAS) and brief pain inventory, vital signs were assessed as well. M technique hand massage was done on both hands and arms for 10 minutes using odourless baby oil, afterwards pain level was re-assessed using usual analogue scale and vital signs were re-evaluated within 10-15 minutes after the completion of the intervention.

In the control group, patient information form was filled, pain level was assessed via visual analogue scale (VAS) and brief pain inventory, vital signs were assessed after obtaining verbal and written consent from the elderly participants. No intervention was done by the researcher for this group except routine treatment, within 10-15 minutes pain level was reassessed using VAS and vital signs were re-evaluated.

Application: aromatherapy is a natural and gentle form of treatment that can access the human body through inhaled scent molecules that activate the limbic system, an area in the brain that plays an important role for emotion and behaviour. It can also be applied as a topical massage which gives soothing and relaxing feeling by stimulating the nervous system that regulates heart rate, blood pressure, stress and breathing patterns. On top of all the benefits, easy application, low cost and low side effects are some of the reasons aromatherapy is accepted as complementary and integrative medicine. M technique hand massage is a unique choreographed method that follows certain type of movement, pressure and pace which is custom made for the most fragile patient. Combining aromatherapy with the M technique hand massage, can give satisfactory results, as this massage technique is an extremely soft, comfortable and relaxing massage type that can be applied to even the most fragile patient.

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of 65 years and older
* who had chronic non-malignant pain for at least three months
* those who had agreed to participate in research
* those who do not have cognitive impairment and can answer questions

Exclusion Criteria:

* patients with dermatological problems on the hand or arm,
* Any swelling or signs of inflammation in the hand or arm,
* those who have neuropathy or loss of sensation in the hand or arm,
* those who have hand deformity,
* those who are allergic to lavender, perfumes or cosmetics,
* those who had undergone Surgery in the last month or so
* those who are diagnosed with Cancer

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 15 minutes
  The visual analogue scale (VAS) is a subjective measure for the level of pain consisting of 10cm horizontal or vertical line, with "0" indicating no pain at one end while "10" indicates very severe pain at the other end. Patients mark the point that corresponds to the pain he/she was experiencing during the interview. The scale was used in this study to evaluate level of chronic pain. This scale is a very sensitive method that helps to evaluate pharmacological and non-pharmacological treatments that reduce pain (Uyar & Yıldırım, 2010).
Brief pain inventor | base line
  Wisconsin Short Pain inventory was developed to evaluate pain status of individuals with cancer or chronic diseases. It consists of 15 items and each item takes a value between 0-10. The lowest score obtained from the brief pain inventory indicates that there is no pain in the last 24 hours, 1-3 points indicate mild pain in the last 24 hours, 4-7 points indicate moderate pain in the last 24 hours, and 8-10 points indicate severe pain in the last 24 hours. The validity and reliability study of the brief pain inventory for patients with chronic non-malignant pain in Turkey was conducted by Yıldırım et al. (2019).
Patient information form | base line
  The individual identiﬁcation form was created by the researchers in the light of information collected from the literature. It was divided into 3 different parts; the ﬁrst part contained sociodemographic characteristics such as age, gender, educational status, occupation, social security, marital status, and number of children. The second part was regarding health-related characteristics such as duration of chronic pain diagnosis whether or not it had been treated, what treatment modality was applied, how long the pain complaint had lasted, the presence of other accompanying illnesses, and general state of health.
Blood Pressure | 15 minutes
  Systolic and diastolic blood pressure was measured with Omron digital arm meter sphygmomanometer.
Pulse Rate | 15 minutes
  Puls rate was counted and evaluated for one whole minute.
Respiratory Rate | 15 minutes
  Respiratory rate was counted and evaluated for one whole minute.
Body Temperature | 15 minutes
  Body temperature was recorded using infrared thermometer.

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Uyar, Professor, Study Director — Ege Unversity; yasemin Yildirim, Professor, Study Director — Ege Unversity; Haben Tesfu Gebreselassie, Study Director — Ege Unversity
Locations (1):
- Ege Unversity Algology polyclinic, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
no planning

DOCUMENTS (1):
  • Study Protocol (2021-02-27): https://cdn.clinicaltrials.gov/large-docs/88/NCT04786288/Prot_000.pdf